CLINICAL TRIAL: NCT06027476
Title: Prognostic Significance of Preoperative Inflammatory Status for Postoperative Acute Kidney Injury in Elderly Patients Undergoing Non-cardiac Surgery
Brief Title: Preoperative Inflammatory Status and Postoperative Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Rao Sun (Other)
Responsible Party: Sponsor-Investigator, Rao Sun, Associate chief physician, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJH-20230608B
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute kidney injury (AKI) is a common complication during the early postoperative period after noncardiac surgery. Patients with AKI are at an increased risk of developing chronic kidney disease, prolonging hospitalization, and experiencing higher rates of morbidity and mortality. Identifying preoperative risk factors for postoperative AKI can significantly contribute to the development of preventive strategies and improved perioperative care in this vulnerable patient population.

The goal of this retrospective study is to investigate the predictive value of preoperative inflammatory status, as measured by complete blood count-derived inflammatory markers, such as the neutrophil-to-lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR), monocyte-to-lymphocyte ratio (MLR), derived neutrophil-to-lymphocyte ratio (dNLR), neutrophil-to-lymphocyte*platelet ratio (NLPR), systemic immune-inflammatory index (SII), systemic inflammatory response index (SIRI), and aggregate index of systemic inflammation (AISI), on postoperative AKI in elderly patients undergoing non-cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥ 65 years.
2. general, gynaecological, neurosurgery, orthopaedic, or thoracic surgery.
3. surgery duration lasting longer than one hour.

Exclusion Criteria:

1. patients with an American Society of Anesthesiologists (ASA) physical status V.
2. those with concurrent cardiac, vascular, transplant or urological surgeries.
3. those with end-stage renal disease (i.e. a glomerular filtration rate of 15 mL/min/1.73 m2 or receiving haemodialysis) or a history of kidney transplantation..
4. those did not have sufficient data required for calculation for inflammatory markers or AKI evaluation.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients (aged ≥ 65 years) who underwent a non-cardiac surgery at Tongji Hospital between July 2018 and December 2021 were included in our study.
Sampling Method: Non-Probability Sample
Enrollment: 8472 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with acute kidney injury after surgery | Within 7 days after surgery
  In accordance with the KDIGO creatinine criteria: a serum creatinine increases of 26.5 mmol/L within 48 hours or 1.5 times baseline within 7 days after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Rao Sun, Wuhan, China

IPD SHARING:
Plan to Share IPD: No